Cover letter

Study protocol

**ORIGINAL TITEL:** 

Comparison between the caudal block and other methods of postoperative pain relief in children undergoing circumcision: A prospective randomized study

Institution review board number (IRB number: 70130623).

**Approval date 13\06\2023** 

The study conforms to the provisions of the Declaration of Helsinki in 1995 (as revised in Edinburgh 2000) and it was ethically approved by the Research Committee for Government Hospitals, Salmaniya Medical Complex, Kingdom of Bahrain (IRB number: 70130623). Selecting the best analgesia method in pediatrics is so important. This is a randomized a prospective study conducted on 90 children who underwent circumcision. The results showed that circumcision in pediatrics using a caudal block can provide longer analgesia for the patient.

ABSTRACT

Background:

Caudal block (CB), dorsal nerve penile block (DPNB), and systemic opioids are common techniques used in pediatric surgeries to provide analgesia for penile surgery such as circumcision.

Aims: This study aimed to compare the effectiveness of the CB with other methods of postoperative pain release.

Material and Methods: The main operation pediatric theater and post-anesthesia recovery unit (PACU) in the Government Hospitals, Salmaniya Medical Complex, Bahrain.

Study subjects: Successive children aged 3 months to 3 years who had American Society of Anesthesiologists with Physical Status classification one and who had undergone elective circumcision

surgery were recruited., Children were randomized to one of three modalities of intraoperative analgesia: CB, or DPNB. And systemic opioids.

study design: Prospective, Observation-randomized, case-controlled trial study. a study Sample size: all patients, for a total of 90 boys going for circumcision surgery. I was recruited over the course of four months, starting in May 2023. The patients will be divided into three groups: A (CB), B systemic opioids, and C (DPsNB). All patients had operations and were observed, and the three groups were compared based on hemodynamic stability, pain scores, duration of sedation,

analgesia need, and parental satisfaction. where the Face, Leg, Activity, and Cry Consolability s(FLACC) pain scale and behaviors were used to observe and compare the three Groups.